29-09-2022

## INFORMED CONSENT

## Searching for meaning;

A study examining the effect of meaning-centered intervention

(PSY-2223-S-0010)

I have read the study information. I have had the opportunity to ask questions about the study (via email), and the questions that I had were answered to my satisfaction.

I had a sufficient amount of time to decide whether I wanted to participate or not.

I understand that the time investment in the current study is substantial (primarily if I am assigned to the treatment group) and stretches out over 10 weeks.

I understand that I am not permitted to participate if I am currently in treatment for an eating disorder or if I am a non-fluent speaker of the English language.

- I voluntarily give informed consent for participation in this study
- In addition, I voluntarily consent to my data being used for the purposes described in the study information. My privacy will be warranted at all times.

If I decide to end my participation, I can do so without providing a reason. If I quit, I will be provided with the opportunity to have my personal data be erased. Once the data is processed and published, it is no longer possible to have your data erased.

| Consent to participate in the research: |
|---|
| [] Yes, I consent to participate. |
| [] No, I do not consent to participate. |
| Consent to processing my personal data: |
| [] Yes, I consent to the processing of my personal data for educational and scientific |
| purposes as mentioned in the research information. I know that one month after my |
| last assessment I can ask to have my data withdrawn and erased. I can also ask for |
| this if I decide to stop participating in the research. |
| [] No, I do not consent to the processing of my personal data. |